CLINICAL TRIAL: NCT04320472
Title: Outcomes in Patients With Acute Encephalopathy and SARS-Cov-2 Infection
Brief Title: Acute Encephalopathy in Critically Ill Patients With COVID-19
Acronym: NeuroCOVID19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ictal Group (Other)
Responsible Party: Sponsor
Other Study IDs: Neuro-COVID-19
Record Dates: First submitted 2020-03-22; First posted 2020-03-25 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: COVID-19; Encephalopathy; Critically Ill
MeSH Terms: conditions — COVID-19; Brain Diseases; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follow up: Follow up of all included patients up to 3 months after enrollement
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — Follow up up to day 90 (Glasgow outcome scale, Glasgow outcome scale extended, functionnal impairments : Barthel index, Disability Rating Scale)

SUMMARY:
Infection with SARS-CoV-2 or severe acute respiratory syndrome coronarvirus type 2 was highlighted in December 2019 in the city of Wuhan in China, responsible for an pandemic evolution since March 11, 2020. The infection affects all ages of life, although affecting children in a very small proportion of cases. The typical presentation of the disease combines fever (98%), cough (76%), myalgia and asthenia (18%) as well as leukopenia (25%) and lymphopenia (63%). Upper airway involvement rare.

The main clinical presentation requiring hospitalization of infected patients is that of atypical pneumonia which may require critical care management (27%), and progress to an acute respiratory distress syndrome (67%) involving life-threatening conditions in almost 25% of patients diagnosed with SARS-CoV-2 infection. Other organ damage have been reported, mainly concerning kidney damage (29%) which may require renal replacement therapy in approximately 17% of patients.

Neurological damage has been very rarely studied, yet reported in 36% of cases in a study including patients of varying severity.

Finally, the mortality associated with this emerging virus is high in patients for whom critical care management is necessary, reported in 62% of patients.

We therefore propose a prospective observational study which aim at reporting the prevalence of acute encephalopathy at initial management in Critical/Intensive care or Neurocritical care , to report its morbidity and mortality and to identify prognostic factors.

DETAILED DESCRIPTION:
All patients with SARS-CoV-2 infection and acute encephalopathy at presentation will be prospectively included in the NEURO-COVD-19 study. This study will collect demographic data, clinical examen at prehospital/emergency room and ICU admission (including neurological signs), and all ancillary exams performed to identify a cause of neurological impairment. Outcome will be evaluated using the Glasgow Outcome Scale score at ICU and hospital discharge, and day-90 after ICU admission.

Acute encephalopathy will be defined as recently stated :

"1. The term acute encephalopathy refers to a rapidly developing (over less than 4 weeks, but usually within hours to a few days) pathobiological process in the brain. This is a preferred term 2. Acute encephalopathy can lead to a clinical presentation of subsyndromal delirium, delirium, or in case of a severely decreased level of consciousness, coma; all representing a change from baseline cognitive status 3. The term delirium refers to a clinical state characterized by a combination of features defined by diagnostic systems such as the DSM-5. Delirium according to the DSM-5 is defined if criterium A-E are fulfilled: A. Disturbance in attention (i.e., reduced ability to direct, focus, sustain, and shift attention) and awareness (reduced orientation to the environment). B. The disturbance develops over a short period of time (usually hours to a few days) represents a change from baseline attention and awareness, and tends to fluctuate in severity during the course of the day. C. An additional disturbance in cognition (e.g., memory deficit, disorientation, language, visuospatial ability, or perception). D. The disturbances in criteria A and C are not explained by another pre-existing, established, or evolving neurocognitive disorder, and do not occur in the context of a severely reduced level of arousal, such as coma. E. There is evidence from the history, physical examination, or laboratory findings that the disturbance is a direct physiologic consequence of another medical condition, substance intoxication or withdrawal (i.e. because of a drug of abuse medication), or exposure to a toxin, or is because of multiple etiologies. " (Slooter, A.J.C., Otte, W.M., Devlin, J.W. et al. Updated nomenclature of delirium and acute encephalopathy: statement of ten Societies. Intensive Care Med (2020). https://doi.org/10.1007/s00134-019-05907-4)

ELIGIBILITY:
Inclusion Criteria:

* Critical/Intensive care or Neurocritical care admission
* Admission for/with acute encephalopathy defined as a rapidly developing (over less than 4 weeks, but usually within hours to a few days) pathobiological process in the brain; including delirium or subsyndromal (DSM V definition) or coma (Glasgow coma scale score < 9)
* SARS-COV-2 infection (respiratory or other PCR specimen)
* Age ≥ 18 years

Exclusion Criteria:

- Opposition to study participation from the patient itself or patient surrogate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute encephalopathy and ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence | at Critical/Intensive care or Neurocritical care admission
  ratio of patients with acute encephalopathy among the total of patients with SARS-Cov-2 infection at Critical/Intensive care or Neurocritical care admission

SECONDARY OUTCOMES:
Favorable outcome | 3 months
  A favorable outcome is defined by a Glasgow Outcome Scale (GOS) of 5. The Glasgow Outcome Scale (GOS) will be determined patients charts review, phone call, and/or general practitioner interview conducted by an independent assessor. The GOS score : [1: Death, 2: Persistent vegetative state, 3: Severe disability, 4: Moderate disability, 5 : Low disability]
Favorable outcome | 3 months
  A favorable outcome is defined by a Glasgow Outcome Scale Extended (GOSe) >= 5. The Glasgow Outcome Scale Extended (GOSe) will be determined patients charts review, phone call, and/or general practitioner interview conducted by an independent assessor. The GOSe score : [1: Death, 2: Persistent vegetative state, 3: Severe disability Lower, 4: Severe disability Upper, 5: Moderate disability Lower, 6: Moderate disability Upper, 7 : Good recovery lower, 8 : Good recovery Upper]

CONTACTS AND LOCATIONS:
Overall Officials: Stephane LEGRIEL, MD, PhD, Principal Investigator — Ictal Group
Locations (39):
- United States (2):
  - Jackson Memorial Health System; University of Miami, Miller School of Medicine, Miami, Florida
  - Wellstar Atlanta Medical Center, Atlanta, Georgia
- Universidade Federal de São Paulo, São Paulo, Brazil
- Fundación Valle del Lili, University Hospital, Cali, Colombia
- Cairo University Hospitals, Cairo, Egypt
- France (32):
  - Centre Hospitalier d'Argenteuil, Argenteuil
  - Centre Hospitalier de Beauvais, Beauvais
  - Centre Hospitalier Universitaire Ambroise Paré, Boulogne
  - Centre Hospitalier de Bourg en Bresse, Bourg-en-Bresse
  - Centre Hospitalier Régional Universitaire de Brest, Brest
  - Centre Hospitalier de Brives, Brive-la-Gaillarde
  - Centre Hospitalier Universitaire Beaujon, Clichy
  - Centre Hospitalier Universitaire Louis Mourier, Colombes
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre hospitalier de Dieppe, Dieppe
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier d'Etampes, Étampes
  - Grand Hôpital de l'Est Francilien - Site de Marne-la-Vallée, Jossigny
  - Centre Hospitalier de la Roche-sur-Yon, La Roche-sur-Yon
  - Centre Hospitalier de La Rochelle, La Rochelle
  - Centre Hospitalier de Versailles, Le Chesnay
  - Centre Hospitalier Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire Hôpital Edouard Herriot, Lyon
  - Hôpital privé Jacques Cartier, Massy
  - Groupe Hospitalier Sud Ile-de-France, Melun
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Centre Hospitalier Universitaire Cochin, Paris
  - Groupe hospitalier Paris Saint-Joseph, Paris
  - Hôpital Fondation Adolphe de Rothschild, Paris
  - Hopital Privé Claude Galien, Quincy-sous-Sénart
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier de Roanne, Roanne
  - Hopital Foch, Suresnes
  - Centre Hospitalier de Toulon, Toulon
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Centre Hospitalier Universitaire de Tours, Tours
  - Gustave-Roussy, Villejuif
- Hospital Regional De Alta Especialidad Del Bajío, Guanajuato City, Mexico
- Hospital Clinic Universitari, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Legriel S, Badenes R, Engrand N, Mendoza-Trujillo R, Soulier P, Benghanem S, Pizzi M, Maciel C, Chelly J, Zuber B, Labruyere M, Plantefeve G, Jacq G, Galbois A, Launey Y, Argaud L, Lesieur O, Ferre A, Paul M, Guillon A, Bailly P, Beuret P, de-Carne MC, Siami S, Benzekri D, Colin G, Gaviria L, Aldana JL, Bruel C, Stoclin A, Sedillot N, Geri G, Samano D, Sobczak E, Swafford E, O'Phelan K, Meffert A, Holleville M, Silva S, Alves da Costa MJ, Mejia J, Alkhachroum A; for NeuroCovid19. Outcomes in Patients With COVID-19 With Acute Encephalopathy and Coma: An International Prospective Study. Neurology. 2023 May 30;100(22):e2247-e2258. doi: 10.1212/WNL.0000000000207263. Epub 2023 Apr 11. PMID 37041081